CLINICAL TRIAL: NCT07261696
Title: The Effects of Inspiratory Muscle Training on the Autonomic Nervous System and Clinical Symptoms in Female Patients With Fibromyalgia
Brief Title: The Effects of Inspiratory Muscle Training Female Patients With Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Gürkan Demirtas, PhD, Nigde Omer Halisdemir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-95860085-050.04-722238
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Fibromyalgia; Autonomic Dysfunction
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group (Experimental): Training at 30% of maximum inspiratory pressure for 6 weeks, 2 sessions per day, 7 days a week
  Interventions: Other: Exercise
- Sham group (Sham Comparator): Training at 0-10% of maximum inspiratory pressure for 6 weeks, 2 sessions per day, 7 days a week
  Interventions: Other: Exercise
- Control group (No Intervention): No Intervention

INTERVENTIONS:
Other: Exercise — Inspiratory muscle training program will be applied to the study and sham group for 7 days/6 weeks.
  Arms: Sham group; Study Group

SUMMARY:
Fibromyalgia is a chronic condition characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and psychological symptoms. Autonomic nervous system (ANS) dysfunction, marked by increased sympathetic and reduced parasympathetic activity, is considered one of its possible mechanisms. Although exercise is recommended in treatment, low motivation and fatigue often limit participation. Therefore, inspiratory muscle training (IMT), which targets the respiratory muscles, is seen as an easy-to-apply alternative.This randomized, controlled, double-blind study will be conducted at Niğde Ömer Halisdemir University Hospital. Fifty-one women aged 18-65 years who meet the 2010/2016 ACR criteria for fibromyalgia will be randomly assigned to three groups: training (30% of maximal inspiratory pressure), sham (0-10%), and control (no training). ANS functions will be assessed using heart rate variability and the COMPASS-31 questionnaire. Pain, sleep quality, fatigue, anxiety, depression, and respiratory muscle strength will also be evaluated. Training will be performed with the Powerbreathe® device twice daily for six weeks.The study aims to investigate the effects of IMT on ANS functions in fibromyalgia and to explore its relationship with symptoms such as pain, fatigue, sleep disturbances, anxiety, and depression.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic disorder characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and psychological symptoms, the exact cause of which remains unclear. Autonomic nervous system (ANS) dysfunction, characterized by increased sympathetic activity and decreased parasympathetic tone, is considered one of the major pathophysiological mechanisms of the disease. Exercise is a strongly recommended non-pharmacological approach in the treatment of fibromyalgia; however, low motivation, fatigue, and poor adherence often limit the applicability of conventional aerobic or resistance exercise programs. Therefore, inspiratory muscle training (IMT), which specifically targets the respiratory muscles, is considered an alternative method that is easy to apply and may have regulatory effects on ANS function.

This randomized, controlled, double-blind, and prospective study will be conducted in the Rheumatology and Cardiology Clinics of Niğde Ömer Halisdemir University Training and Research Hospital. A total of 51 female participants aged 18-65 years who meet the 2010/2016 American College of Rheumatology (ACR) criteria for fibromyalgia will be randomly assigned to three groups: the training group (30% maximal inspiratory pressure [MIP]), the sham group (0-10% MIP), and the control group (no training). ANS functions will be evaluated by heart rate variability (HRV) and the COMPASS-31 questionnaire. Pain will be assessed using the Visual Analog Scale and pressure pain threshold; sleep quality by the Pittsburgh Sleep Quality Index; fatigue by the Modified Fatigue Impact Scale; anxiety and depression by the Hospital Anxiety and Depression Scale; and respiratory muscle strength by the Powerbreathe® K5 device. Training will be performed using the Powerbreathe® Classic device twice daily, seven days per week, for six weeks.

The primary aim of this study is to evaluate the effects of inspiratory muscle training on autonomic nervous system functions in patients with fibromyalgia. Secondarily, the effects of this training on symptoms such as pain, fatigue, sleep disturbances, anxiety, and depression, as well as the relationship between these symptoms and changes in ANS activity, will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 18 and 65 years old,
* Have been diagnosed with fibromyalgia according to the 2010/2016 ACR criteria,
* Be female,
* Have moderate pain lasting at least 3 months and defined as at least 30 mm on the 0-100 mm visual analogue scale (VAS).

Exclusion Criteria:

* Presence of chronic heart disease,
* Current use of narcotic drugs,
* History of asthma or other chronic respiratory diseases,
* Pregnancy,
* Diabetes, kidney, adrenal, pituitary or thyroid disorders,
* History of serious neurological or psychiatric disorders (e.g. mania, psychosis, suicidal tendencies, bipolar disorder, schizophrenia, autism spectrum disorders),
* Neurodegenerative diseases (e.g. Parkinson's, Alzheimer's, Huntington's disease),
* Head trauma, migraine,
* Presence of active cardiac implants.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Autonomic nervous system- HRV | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  The procedure will be performed using a 24-hour ECG Holter monitor.
Autonomic Nervous System- COMPASS-31 | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  The Composite Autonomic Symptom Score-31 questionnaire will be used.

SECONDARY OUTCOMES:
Pain- Visual Analogue Scale | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  Visual Analogue Scale will be used.
Pain- Pressure Pain Treshold | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  The pain threshold will be assessed using a standard pressure algometer
Sleep- Pittsburgh sleep quality index | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  Pittsburgh sleep quality index questionnaire will be used.
Fatigue- Modified Fatigue Impact Scale | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  Modified Fatigue Impact Scale will be used.
Anxiety and Depression- Hospital Anxiety and Depression Scale | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  Hospital Anxiety and Depression Scale questionnaire will be used.
Maximal inspiratory pressure | At the time participants joined the study and after the 6-week training for the intervention and sham groups, and 6 weeks later for the control group.
  Measurements will be taken using the PowerBreathe K5 MIP device to determine the exercise load.

CONTACTS AND LOCATIONS:
Overall Officials: Gürkan Demirtaş, PhD, Principal Investigator — Niğde Ömer Halisdemir University
Locations (1):
- Niğde Ömer Halisdemir Üniversitesi, Niğde, Niğde Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No